CLINICAL TRIAL: NCT03702686
Title: Pilot Study of the FEEDBACK System for Use With Infants in the Neonatal Intensive Care Unit (NICU) at the University of Virginia (UVA)
Brief Title: Pilot Study of the FEEDBACK System for Use With Infants in the Neonatal Intensive Care Unit at University of Virginia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: evaluating feasibility
Sponsor: Molex Ventures LLC (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Prot-01-UVA rev 3
Record Dates: First submitted 2018-10-02; First posted 2018-10-11 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Breastfeeding
Keywords: breastfeeding, pre-term infant, NICU
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FEEDBACK system (Experimental): Mother / infant dyad will use the FEEDBACK system during a breastfeeding session.
  Interventions: Device: FEEDBACK System

INTERVENTIONS:
Device: FEEDBACK System — Smart Nipple Shield and Monitor Unit

SUMMARY:
The purpose of this study is to assess the accuracy of FEEDBACK for measuring breastmilk intake of a pre-term baby. Mothers and babies will use the FEEDBACK system during a breastfeeding session in the NICU. Babies will be weighed prior to breastfeeding and again after breastfeeding. The weight gain of the baby will be compared to the volume measured using FEEDBACK. The study will also evaluate the device safety and ease of use.

DETAILED DESCRIPTION:
Researchers have long stated that accurate assessment of infant milk intake while breastfeeding is needed for clinical practice and research. Many methods for measuring milk intake have been studied. While the intake of formula fed infants can be directly measured based on the amount of fluid in the bottle, determining the actual milk intake for breastfed infants is more difficult. Precise feed volumes are especially important for infants in the NICU. Most premature infants are unable to breastfeed because they are not able to coordinate suckling and swallowing.

The FEEDBACK system includes a nipple shield and a monitoring unit. It helps protect the nipple of a breastfeeding mother as well as measures and displays the volume of milk, in mL or oz, that an infant consumes during a breast feeding session. Based on this information, a mother has quantitative data regarding her infant's milk intake for her own use or to share with her health care provider.

This study is designed in two phases. First, data will be collected from breastfeeding mothers of pre-term infants to develop an algorithm that can identify feeding patterns in the pre-term infant. Once established, accuracy of FEEDBACK will be assessed comparing pre and post weights of the breastfed infant to the volume intake measured by FEEDBACK.

ELIGIBILITY:
Inclusion Criteria:

1. Mother willing and able to provide informed consent for herself and her infant to participate in the study
2. Mother / infant dyad has an indication for and is currently using a nipple shield as per Licensed Independent Practitioner (LIP) or UVA lactation consultant assessment and recommendation.
3. FEEDBACK Smart Nipple Shield 'fit' assessment has been done by a study team member. Size to be comparable to the Smart Nipple Shield sizes (20mm or 24mm)
4. Infant is <37 weeks corrected gestational age at time of first planned FEEDBACK feed and in the NICU
5. Infant must be medically cleared for PO feeding as determined by presence of a milestone feeding order documented in EPIC.
6. Mother willing to be present for PO feeding sessions per study requirements.

Exclusion Criteria:

1. Infant with an oral, pharyngeal or mandibular abnormality where the use of a nipple shield would be contraindicated.
2. Mother / infant dyad deemed ineligible based on LIP or lactation consultant assessment.
3. Mother's with multiples > than 2. For example, if mother has triplets only 2 of the 3 infants are allowed to be in the study.
4. Infant on any isolation precautions.
5. Infant receiving any IV fluids.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of pre and post test weights (grams) during a breastfeeding session compared to the volume calculated by the FEEDBACK system. | 3 weeks per mother / infant dyad; up to 5 feedings
  The weight of the pre-term infant will be measured (grams) before and after breastfeeding. During the feeding the FEEDBACK system records digital signals which are used to calculate flow rate and volume. The weight gain (grams) will then be compared to the volume calculated by FEEDBACK to develop the algorithm.
Accuracy (in grams) of the FEEDBACK system, based on comparison of the pre and post breastfeeding test weights to the calculated FEEDBACK volume. | 2 weeks per mother / infant dyad; 5 feedings
  The weight of the pre-term infant will be measured (grams) before and after breastfeeding. The weight gain will be compared to the FEEDBACK volume to calculate accuracy.

SECONDARY OUTCOMES:
Measure the Device Ease of Use via a questionnaire | 2 weeks, (after feeding session 5) for each mother/infant dyad
  Measure the mother's ease of use for the the FEEDBACK system based on a series of questions with a score of 1 - 5. (1 = difficult, 5 = easy)
Measure the Mother's Perception of Breastfeeding via a questionnaire | 2 weeks, (prior to feeding session 1 and after feeding session 5) for each mother/infant dyad
  Measure the mother's perception of breastfeeding based on a series of questions with a score of 1 - 5 (1 = difficult, 5 = easy) (Pilot Phase)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Vergales, MD, Principal Investigator — University of Virginia, Division of Neonatology, Department of Pediatrics
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States